CLINICAL TRIAL: NCT04233216
Title: A Phase 3, Randomized, Clinical Study in HIV-1-Infected Heavily Treatment-Experienced Participants Evaluating the Antiretroviral Activity of Blinded Islatravir (ISL), Doravirine (DOR), and Doravirine/Islatravir (DOR/ISL), Each Compared to Placebo, and the Antiretroviral Activity, Safety, and Tolerability of Open-Label DOR/ISL
Brief Title: Doravirine/Islatravir (DOR/ISL) in Heavily Treatment-Experienced (HTE) Participants for Human Immunodeficiency Virus Type 1 (HIV-1) Infection (MK-8591A-019)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8591A-019; MK-8591A-019 (Other: MSD); 205243 (Registry Identifier: JAPIC-CTI); 2019-000588-26 (EudraCT Number)
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Results first posted 2023-12-08 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — islatravir; doravirine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ISL + ART (Experimental): HTE participants with HIV-1 infection take ISL 0.75 mg once daily (QD) in combination with failing ART from Day 1 to Day 7; followed by open-label 100 mg DOR/0.75 mg ISL fixed dose combination (FDC) QD + OBT from Day 8 to Week 97.
  Interventions: Drug: ISL; Drug: DOR/ISL
- DOR + ART (Experimental): HTE participants with HIV-1 infection take DOR 100 mg QD in combination with failing ART from Day 1 to Day 7; followed by open-label 100 mg DOR/0.75 mg ISL FDC QD + OBT from Day 8 to Week 97.
  Interventions: Drug: DOR; Drug: DOR/ISL
- DOR/ISL + ART (Experimental): HTE participants with HIV-1 infection take 100 mg DOR/0.75 mg ISL FDC QD in combination with failing ART from Day 1 to Day 7; followed by open-label 100 mg DOR/0.75 mg ISL FDC QD + OBT from Day 8 to Week 97.
  Interventions: Drug: DOR/ISL
- Placebo + ART (Placebo Comparator): HTE participants with HIV-1 infection take placebo QD in combination with failing ART from Day 1 to Day 7; followed by open-label 100 mg DOR/0.75 mg ISL FDC QD + OBT from Day 8 to Week 97.
  Interventions: Drug: DOR/ISL; Drug: Placebo to ISL; Drug: Placebo to DOR

INTERVENTIONS:
Drug: ISL — ISL 0.75 mg capsule taken by mouth.
  Other Names: Islatravir; MK-8591
  Arms: ISL + ART
Drug: DOR — DOR 100 mg tablet taken by mouth.
  Other Names: Doravirine; MK-1439
  Arms: DOR + ART
Drug: DOR/ISL — 100 mg DOR/0.75 mg ISL FDC taken by mouth.
  Other Names: Doravirine/Islatravir; MK-8591A
Drug: Placebo to ISL — Placebo capsule matched to ISL taken by mouth.
  Arms: Placebo + ART
Drug: Placebo to DOR — Placebo tablet matched to DOR taken by mouth.
  Arms: Placebo + ART

SUMMARY:
This is a 2-part, phase 3 clinical study evaluating the antiretroviral activity and safety/tolerability of islatravir (ISL), doravirine (DOR), and a fixed dose combination (FDC) of DOR/ISL (also known as MK-8591A) in heavily treatment-experienced (HTE) participants with human immunodeficiency virus type 1 (HIV-1) infection. It is hypothesized that the percentage of participants receiving DOR/ISL to achieve ≥0.5 log10 decrease in HIV-1 ribonucleic acid (RNA) from study baseline (Day 1) to Day 8 is superior to placebo, each given in combination with failing antiretroviral therapy (ART).

DETAILED DESCRIPTION:
Part 1 of this study (Day 1 to Day 7) is the double-blind period in which participants receive either ISL, DOR, DOR/ISL, or placebo. Part 2 of this study (Day 8 to Week 97) is the open-label period in which all participants receive DOR/ISL + optimized background therapy (OBT).

ELIGIBILITY:
Inclusion Criteria:

* Is HIV-1 positive.
* Has been receiving the same baseline ART for ≥3 months prior to signing the Informed Consent Form/Assent Form.
* Weighs ≥35 kg.
* Has at least triple-class resistance (must include nucleoside reverse transcriptase inhibitor [NRTI], non-nucleoside reverse transcriptase inhibitor [NNRTI], and resistance to either protease inhibitor (PI) or integrase strand transfer inhibitor (InSTI), based on central laboratory-based resistance or proviral DNA resistance testing at the Screening Visit, or historical resistance testing within 12 months of screening.
* Has ≤2 fully active antiretroviral drugs remaining among all antiretroviral classes that can be effectively combined to form a viable regimen based on resistance, tolerability, safety, drug access, or acceptability to participant.
* If female, is not pregnant or breastfeeding, and is: 1) not a woman of childbearing potential (WOCBP); 2) a WOCBP and uses an acceptable method of contraception/is abstinent; or 3) a WOCBP and has a negative pregnancy test within 24 hours of the first dose of study medication.

Exclusion Criteria:

* Has HIV type 2 (HIV-2) infection.
* Has hypersensitivity or other contraindication to any of the components of the study interventions as determined by the investigator.
* Has hepatitis B virus (HBV) co-infection (defined as hepatitis B surface antigen [HBsAg]-positive or HBV deoxyribonucleic acid [DNA] positive) and is not currently being treated for HBV.
* Has a history or current evidence of any condition, therapy (including active TB co-infection), laboratory abnormality or other circumstance (including drug or alcohol abuse or dependence) that might, in the opinion of the investigator, confound the results of the study or interfere with study participation for the full study duration.
* Is taking or is anticipated to require any of the prohibited therapies from the Screening Visit and throughout the study treatment period.
* Is taking DOR as part of his/her current failing antiretroviral regimen.
* Is taking efavirenz (EFV), etravirine, or nevirapine.
* Is currently participating in or has participated in an interventional clinical study with an investigational compound or device from the Screening Visit through the study treatment period.
* Is female and is expecting to conceive or donate eggs at any time during the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (98):
- United States (19):
  - University of Alabama at Birmingham 1917 Research Clinic ( Site 4031), Birmingham, Alabama
  - Men's Health Foundation ( Site 4018), Los Angeles, California
  - Palmtree Clinical Research, Inc. ( Site 4016), Palm Springs, California
  - Yale School of Medicine ( Site 4007), New Haven, Connecticut
  - Georgetown University Hospital ( Site 4015), Washington D.C., District of Columbia
  - The Kinder Medical Group ( Site 4014), Miami, Florida
  - Orlando Immunology Center ( Site 4012), Orlando, Florida
  - Triple O Research Institute, P.A. ( Site 4020), West Palm Beach, Florida
  - Chatham County Health Department ( Site 4029), Savannah, Georgia
  - Howard Brown Health Center ( Site 4006), Chicago, Illinois
  - Northstar Healthcare ( Site 4004), Chicago, Illinois
  - University of Maryland ( Site 4023), Baltimore, Maryland
  - The University of Mississippi Medical Center ( Site 4036), Jackson, Mississippi
  - Saint Michael's Medical Center-Research - Infectious Disease ( Site 4035), Newark, New Jersey
  - Icahn School of Medicine at Mount Sinai ( Site 4000), New York, New York
  - University of North Carolina at Chapel Hill ( Site 4026), Chapel Hill, North Carolina
  - Saint Hope Foundation, Inc. ( Site 4034), Bellaire, Texas
  - North Texas Infectious Diseases Consultants, PA ( Site 4005), Dallas, Texas
  - Dr. Peter Shalit, MD ( Site 4002), Seattle, Washington
- Australia (5):
  - Holdsworth House Medical Practice ( Site 5300), Sydney, New South Wales
  - St Vincent's Hospital ( Site 5309), Sydney, New South Wales
  - Holdsworth House Medical Practice - Brisbane ( Site 5312), Brisbane, Queensland
  - Monash Health-Monash Medical Centre ( Site 5313), Clayton, Victoria
  - The Alfred Hospital ( Site 5304), Melbourne, Victoria
- Canada (5):
  - Vancouver ID Research and Care Centre Society ( Site 4100), Vancouver, British Columbia
  - Hamilton Health Sciences ( Site 4115), Hamilton, Ontario
  - Ottawa Hospital Research Institute ( Site 4111), Ottawa, Ontario
  - Toronto General Hospital - University Health Network ( Site 4105), Toronto, Ontario
  - McGill University Health Center - Research Institute-CVIS Clinical Research Unit ( Site 4102), Montreal, Quebec
- Chile (3):
  - Fundacion Arriaran ( Site 4401), Santiago, Region M. de Santiago
  - Centro Cardiovascular Cardiosur ( Site 4407), Santiago, Region M. de Santiago
  - Hospital Dr. Hernan Henriquez Aravena ( Site 4405), Temuco, Región de la Araucanía
- Colombia (2):
  - Clinica Colsanitas S.A. Sede Clinica Universitaria Colombia ( Site 4306), Bogotá, Bogota D.C.
  - Fundacion Valle del Lili ( Site 4301), Cali, Valle del Cauca Department
- France (11):
  - Hopital Edouard Herriot ( Site 4726), Lyon, Ain
  - A.P.H. Paris. Hopital Bichat Claude Bernard ( Site 4724), Paris, Ain
  - CHU de Nice Hopital Archet 1 ( Site 4703), Nice, Alpes-Maritimes
  - Hopital Europeen Marseille ( Site 4717), Marseille, Bouches-du-Rhone
  - CHU de Bordeaux- Hopital Saint Andre ( Site 4715), Bordeaux, Gironde
  - CHU de Rouen ( Site 4705), Rouen, Haute-Normandie
  - CHU de Montpellier - Hopital Saint-Eloi ( Site 4721), Montpellier, Herault
  - Centre Hospitalier de Tourcoing ( Site 4700), Tourcoing, Nord
  - Hopital Avicenne ( Site 4702), Bobigny, Seine-Saint-Denis
  - Hopital Hotel Dieu [Paris, France] ( Site 4723), Paris
  - A.P.H. Paris, Hopital Saint Louis ( Site 4714), Paris
- Germany (6):
  - Medizinische Hochschule Hannover ( Site 4612), Hanover, Lower Saxony
  - Universitaetsklinikum Bonn ( Site 4600), Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Essen ( Site 4607), Essen, North Rhine-Westphalia
  - ZIBP-Zentrum fur Infektiologie Berlin Prenzlauer Berg GmbH ( Site 4603), Berlin
  - EPIMED GmbH ( Site 4608), Berlin
  - ICH Study Center GmbH & Co.KG ( Site 4609), Hamburg
- Italy (9):
  - Azienda Ospedaliero Universitaria di Modena Policlinico ( Site 5004), Modena, Emilia-Romagna
  - Ospedale San Gerardo ASST Monza ( Site 5012), Monza, Monza E Brianza
  - Fondazione IRCCS Ca' Granda-Ospedale Maggiore Policlinico ( Site 5001), Milan
  - Universita' Vita Salute. Ospedale San Raffaele ( Site 5002), Milan
  - Azienda Ospedaliera San Paolo ( Site 5003), Milan
  - ASST Fatebenefratelli-Ospedale Sacco ( Site 5000), Milan
  - IRCCS Policlinico San Matteo ( Site 5010), Pavia
  - Istituto Nazionale per Le Malattie Infettive Lazzaro Spallanzani ( Site 5005), Roma
  - Policlinico Gemelli Instituto di Clinica Chirurgica ( Site 5006), Roma
- Center Hospital of the National Center for Global Health and Medicine ( Site 5401), Tokyo, Japan
- Peru (3):
  - INMENSA ( Site 4506), Lima, Muni Metro de Lima
  - Via Libre ( Site 4500), Lima
  - Policlinico Universidad Nacional Mayor de San Marcos ( Site 4501), Lima
- Portugal (5):
  - Hospital de Nossa Senhora da Oliveira- EPE ( Site 4905), Guimarães, Braga District
  - Hospital Dr. Fernando Fonseca, EPE - Amadora/Sintra ( Site 4902), Amadora, Lisbon District
  - Centro Hospitalar de Lisboa Norte Hospital de Santa Maria ( Site 4913), Lisbon
  - Hospital Geral de Santo Antonio ( Site 4908), Porto
  - Centro Hospitalar de Sao Joao. EPE - Hospital de Sao Joao ( Site 4907), Porto
- HOPE Clinical Research ( Site 5700), San Juan, Puerto Rico
- Russia (7):
  - Saint Petersburg Center for Prophylactic of AIDS and Inf. Diseases ( Site 5101), Saint Petersburg, Leningradskaya Oblast'
  - Infectious Clinical Hospital #2 ( Site 5114), Moscow, Moscow
  - Gbuz Samarskiy Oblastnoy Klinicheskiy Tsentr Profilaktiki I Bor'by So Spid ( Site 5113), Samara, Samara Oblast
  - FGU Republican Clinical Infectious Hospital of Roszdrav ( Site 5100), Saint Petersburg, Sankt-Peterburg
  - Smolensk Center On Aids And Infectious Diseases Prophylaxis ( Site 5115), Smolensk, Smolensk Oblast
  - Regional Center for Prevent. and Control of AIDS and Inf. Diseases ( Site 5106), Yekaterinburg, Sverdlovsk Oblast
  - Republican Clinical Hospital of Infectious Diseases n. a. A.F.Agafonov ( Site 5104), Kazan', Tatarstan, Respublika
- South Africa (4):
  - FARMOVS ( Site 4805), Bloemfontein, Free State
  - Wits Clinical HIV Research Unit ( Site 4804), Johannesburg, Gauteng
  - Ezintsha ( Site 4806), Johannesburg, Gauteng
  - King Edward Hospital ( Site 4802), Durban, KwaZulu-Natal
- South Korea (3):
  - Pusan National University Hospital ( Site 5503), Busan, Pusan-Kwangyokshi
  - Severance Hospital Yonsei University Health System ( Site 5500), Seoul
  - The Catholic University of Korea. Seoul St. Mary s Hospital ( Site 5502), Seoul
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol ( Site 5600), Badalona, Barcelona
  - Hospital Clinic i Provincial ( Site 5601), Barcelona, Catalonia
  - Hospital Santa Lucia ( Site 5603), Cartagena, Murcia, Region de
  - Hospital Universitario La Paz ( Site 5604), Madrid
- Ukraine (8):
  - Dnipropetrovsk Regional Center of Socially Significant Diseases ( Site 5619), Dnipro, Dnipropetrovsk Oblast
  - Regional Clinical Infectious Hospital ( Site 5614), Kharkiv, Kharkivs’ka Oblast’
  - Kherson City Clinical Hospital n.a. Y.Y. Karabelesh ( Site 5620), Kherson, Kherson Oblast
  - Institute of Epidemiology and Infect Diseases of the NAMS of Ukraine ( Site 5615), Kyiv, Kyivska Oblast
  - Mykolaiv center of paliative assistance and integrated services ( Site 5621), Mykolayiv, Mykolaiv Oblast
  - MNE Odesa Regional Center of Socially Significant Diseases ( Site 5611), Odesa, Odesa Oblast
  - MI Vinnytsia Regional Center of AIDS Prevention and Care ( Site 5618), Berezina, Vinnytsia Oblast
  - Kyiv City Clinical Hospital 5 ( Site 5616), Kyiv
- United Kingdom (2):
  - Royal Free Hospital ( Site 5202), London, Camden
  - Western General Hospital ( Site 5201), Edinburgh, Edinburgh, City of

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Carr A, Mngqibisa R, Khaertynova I, Kumar PN, Haider S, Zhang Y, Correll T, Asante-Appiah E, Greaves W. Efficacy and safety of doravirine/islatravir in heavily treatment-experienced participants living with HIV-1: results from a randomized trial. AIDS. 2026 Feb 1;40(2):189-197. doi: 10.1097/QAD.0000000000004367. Epub 2025 Oct 1. PMID 41037024
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26356&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Heavily Treatment-Experienced (HTE) adult participants with Human Immunodeficiency Virus Type 1 (HIV-1) infection and currently on failing antiretroviral therapy (ART) were enrolled in this study.
Groups:
- ISL + ART: HTE participants with HIV-1 infection took islatravir (ISL) 0.75 mg once daily (QD) in combination with failing ART from Day 1 to Day 7; followed by open-label 100 mg doravirine (DOR)/0.75 mg ISL fixed dose combination (FDC) QD + optimized background therapy (OBT) from Day 8 to Week 97.
- DOR + ART: HTE participants with HIV-1 infection took DOR 100 mg QD in combination with failing ART from Day 1 to Day 7; followed by open-label 100 mg DOR/0.75 mg ISL FDC QD + OBT from Day 8 to Week 97.
- DOR/ISL + ART: HTE participants with HIV-1 infection took 100 mg DOR/0.75 mg ISL FDC QD in combination with failing ART from Day 1 to Day 7; followed by open-label 100 mg DOR/0.75 mg ISL FDC QD + OBT from Day 8 to Week 97.
- Placebo + ART: HTE participants with HIV-1 infection took placebo QD in combination with failing ART from Day 1 to Day 7; followed by open-label 100 mg DOR/0.75 mg ISL FDC QD + OBT from Day 8 to Week 97.
Period: Overall Study
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Started | 7 | 14 | 7 | 7
Completed | 6 | 9 | 4 | 5
Not Completed | 1 | 5 | 3 | 2
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 3 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- ISL + ART: HTE participants with HIV-1 infection took ISL 0.75 mg once daily (QD) in combination with failing ART from Day 1 to Day 7; followed by open-label 100 mg DOR/0.75 mg ISL fixed dose combination (FDC) QD + OBT from Day 8 to Week 97.
- Total: Total of all reporting groups
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART | Total
Number analyzed (Participants) | 7 | 14 | 7 | 7 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (12.7) | 48.6 (11.8) | 54.0 (10.0) | 44.6 (9.1) | 48.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 1 | 8
  Male | 5 | 10 | 6 | 6 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 0 | 4
  Not Hispanic or Latino | 7 | 12 | 5 | 7 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 0 | 1 | 11
  White | 2 | 7 | 6 | 5 | 20
  More than one race | 0 | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Plasma HIV-1 RNA [Mean (Standard Deviation); unit: Log10 copies/mL] | 4.1 (0.8) | 4.3 (0.9) | 4.5 (0.8) | 4.2 (0.7) | 4.3 (0.8)
Custer of differentiation 4+ (CD4+) T-cell Count [Mean (Standard Deviation); unit: cells/mm^3] | 166.3 (121.7) | 132.4 (136.6) | 178.6 (135.5) | 132.6 (100.7) | 148.5 (123.3)
Genotypic resistance [Count of Participants; unit: Participants]
  Nucleos(t)ide reverse transcriptase inhibitor (NRTI) substitutions | 7 | 14 | 7 | 7 | 35
  Non-nucleoside reverse transcriptase inhibitor (NNRTI) substitutions | 7 | 14 | 7 | 7 | 35
  Protease inhibitor (PI) substitutions | 7 | 14 | 7 | 7 | 35
  Integrase strand transfer inhibitor (InSTI )substitutions | 5 | 9 | 5 | 6 | 25
Phenotypic resistance [Count of Participants; unit: Participants]
  NRTI | 7 | 14 | 7 | 7 | 35
  NNRTI | 6 | 13 | 7 | 7 | 33
  PI | 7 | 12 | 7 | 6 | 32
  InSTI | 5 | 9 | 5 | 7 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Receiving Doravirine/Islatravir (DOR/ISL) With ≥0.5 log10 Change From Day 1 Baseline to Day 8 in Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) Compared to Placebo Treatment
Description: Participants with a ≥0.5 log10 decrease from Day 1 baseline to Day 8 in HIV-1 RNA were identified by the central laboratory with an Abbott Real Time Polymerase Chain Reaction (PCR) assay which has a lower limit of detection (LLOD) of 40 copies/mL Only participants treated with DOR/ISL FDC or placebo were analyzed in this outcome measure.
Time Frame: Day 1 (baseline) and Day 8
Population: All randomized participants who received at least 1 dose of study intervention based on the treatment group to which they were randomized and had baseline data for those analyses that require baseline data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 0 | 0 | 7 | 7
Percentage of participants |  |  | 85.7 [42.1 to 99.6] | 0.0 [0.0 to 41.0]

2. Primary Outcome: Percentage of Participants With ≥1 AEs Through Week 49
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 49 weeks
Population: All randomized participants who received at least 1 dose of study intervention based on the treatment group to which they were randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 7 | 7
Percentage of participants | 71.4 | 85.7 | 85.7 | 85.7

3. Primary Outcome: Percentage of Participants Withdrawing From Study Treatment Due to AE(s) Through Week 25
Description: as for outcome 2
Time Frame: Up to 25 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 7 | 7
Percentage of participants | 0.0 | 7.1 | 14.3 | 0.0

4. Primary Outcome: Percentage of Participants With ≥1 Adverse Events (AEs) Through Week 25
Description: as for outcome 2
Time Frame: Up to 25 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 7 | 7
Percentage of participants | 42.9 | 85.7 | 85.7 | 85.7

5. Primary Outcome: Percentage of Participants Withdrawing From Study Treatment Due to AE(s) Through Week 49
Description: as for outcome 2
Time Frame: Up to 49 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 7 | 7
Percentage of participants | 0.0 | 14.3 | 14.3 | 0.0

6. Secondary Outcome: Percentage of Participants With ≥1 Adverse Events (AEs) Through Week 97
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 97 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 7 | 7
Percentage of participants | 85.7 | 100.0 | 85.7 | 100.0

7. Secondary Outcome: Percentage of Participants Discontinuing From Study Therapy Due to AE(s) Through Week 97
Description: as for outcome 6
Time Frame: Up to 97 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 7 | 7
Percentage of participants | 0.0 | 21.4 | 28.6 | 14.3

8. Secondary Outcome: Percentage of Participants Receiving DOR or ISL (Given With Antiretroviral Therapy [ART]) With ≥0.5 log10 Change From Day 1 Baseline to Day 8 HIV-1 RNA Compared to Placebo Treatment
Description: Participants with a ≥0.5 log10 decrease from Day 1 baseline to Day 8 in HIV-1 RNA were identified by the central laboratory with an Abbott Real Time PCR assay which has a LLOD of 40 copies/mL Only participants treated with either DOR or ISL or placebo (given with ART) were analyzed in this outcome measure. Participants treated with DOR/ISL FDC were not analyzed in this outcome measure.
Time Frame: Day 1 (baseline) and Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 0 | 7
Percentage of participants | 28.6 [3.7 to 71.0] | 78.6 [49.2 to 95.3] |  | 0.0 [0.0 to 41.0]

9. Secondary Outcome: Mean Change From Baseline Day 1 to Day 8 in HIV-1 RNA Following Treatment With DOR/ISL (Given With ART), DOR, or ISL Compared to Placebo Treatment
Description: The change from baseline Day to Day 8 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% confidence intervals (CIs) were calculated based on the t-distribution.
Time Frame: Day 1 (baseline) and Day 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Log10 Copies/mL
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 7 | 7
Log10 Copies/mL | -0.44 [-0.96 to 0.07] | -0.96 [-1.38 to -0.54] | -1.23 [-1.72 to -0.75] | 0.03 [-0.15 to 0.21]

10. Secondary Outcome: Percentage of Participants Receiving DOR/ISL (Given With ART), DOR, or ISL With ≥1.0 log10 Change From Day 1 Baseline to Day 8 HIV-1 RNA Compared to Placebo Treatment
Description: Participants with a ≥1.0 log10 decrease from baseline (Day 1) to Day 8 in HIV-1 RNA were identified by at the central laboratory with an Abbott Real Time Polymerase Chain Reaction (PCR) assay which has a LLOD of 40 copies/mL
Time Frame: Day 1 (baseline) and Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 7 | 7
Percentage of participants | 14.3 [0.4 to 57.9] | 50.0 [23.0 to 77.0] | 85.7 [42.1 to 99.6] | 0.0 [0.0 to 41.0]

11. Secondary Outcome: Percentage of Participants Receiving DOR/ISL (Given With ART) With ≥0.5 log10 Change From Day 1 Baseline to Day 8 in HIV-1 RNA Compared to DOR or ISL Treatment
Description: Participants with a ≥0.5 log10 decrease from baseline (Day 1) to Day 8 in HIV-1 RNA were identified by at the central laboratory with an Abbott Real Time PCR assay which has a lower limit of detection (LLOD) of 40 copies/mL Only participants treated with DOR/ISL or DOR alone or ISL alone were analyzed in this outcome measure. Participants treated with placebo were not analyzed in this outcome measure.
Time Frame: Day 1 (baseline) and Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 7 | 0
Percentage of participants | 28.6 [3.7 to 71.0] | 78.6 [49.2 to 95.3] | 85.7 [42.1 to 99.6] |

12. Secondary Outcome: Mean Change From Baseline Day 1 to Day 8 in HIV-1 RNA Following Treatment With DOR/ISL (Given With ART) Compared to DOR or ISL Treatment
Description: The change from baseline Day 1 to Day 8in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% CIs were calculated based on the t-distribution. The group treated with placebo were not analyzed in this outcome measure.
Time Frame: Day 1 (baseline) and Day 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Log10 Copies/mL
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 7 | 0
Log10 Copies/mL | -0.44 [-0.96 to 0.07] | -0.96 [-1.38 to -0.54] | -1.23 [-1.72 to -0.75] |

13. Secondary Outcome: Percentage of Participants Receiving DOR/ISL (Given With ART) With ≥1.0 log10 Change From Day 1 Baseline to Day 8 in HIV-1 RNA Compared to DOR or ISL Treatment
Description: Participants receiving DOR/ISL with a ≥1.0 log10 decrease from baseline (Day 1) to Day 8 in HIV-1 RNA were identified by at the central laboratory with an Abbott Real Time PCR assay which has a lower limit of detection (LLOD) of 40 copies/mL Only participants treated with DOR/ISL or DOR alone or ISL alone were analyzed in this outcome measure. Participants treated with placebo were not analyzed in this outcome measure.
Time Frame: Day 1 (baseline) and Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 7 | 0
Percentage of participants | 14.3 [0.4 to 57.9] | 50.0 [23.0 to 77.0] | 85.7 [42.1 to 99.6] |

14. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With ≥0.5 log10 Change From Day 1 Baseline to Week 25 in HIV-1 RNA
Description: The percentage of participants in the pooled treatment group with ≥0.5 log10 change from baseline Day 1 to Week 25 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 1 (baseline) and Week 25
Population: Randomized participants who received at least 1 dose of study intervention, had baseline data for those analyses that require baseline data, and had not committed any major protocol violations. Examples of protocol violations include, but are not limited to nonadherence to study intervention; or becoming pregnant.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pooled Treatment: HTE participants with HIV-1 infection from the original four treatment groups (DOR, ISL, DOR/ISL FDC, placebo QD) treated in combination with failing ART from Day 1 to Day 7; followed by treatment with open-label 100 mg DOR/0.75 mg ISL FDC QD + OBT from Day 8 to Week 97 were pooled into a single group as planned per protocol
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 34
Percentage of participants | 85.3 [68.9 to 95.0]

15. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With ≥0.5 log10 Change From Day 1 Baseline to Week 49 in HIV-1 RNA
Description: The percentage of participants in the pooled treatment group with ≥0.5 log10 change from baseline Day 1 to Week 49 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 1 (baseline) and Week 49
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 31
Percentage of participants | 80.6 [62.5 to 92.5]

16. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With ≥0.5 log10 Change From Day 1 Baseline to Week 97 in HIV-1 RNA
Description: The percentage of participants in the pooled treatment group with ≥0.5 log10 change from baseline Day 1 to Week 97 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 1 (baseline) and Week 97
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 26
Percentage of participants | 84.6 [65.1 to 95.6]

17. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With ≥0.5 log10 Change From Day 8 Baseline to Week 25 in HIV-1 RNA
Description: The percentage of participants in the pooled treatment group with ≥0.5 log10 change from baseline Day 8 to Week 25 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 8 (baseline) and Week 25
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 34
Percentage of participants | 64.7 [46.5 to 80.3]

18. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With ≥0.5 log10 Change From Day 8 Baseline to Week 49 in HIV-1 RNA
Description: The percentage of participants in the pooled treatment group with ≥0.5 log10 change from baseline Day 8 to Week 49 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 8 (baseline) and Week 49
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 31
Percentage of participants | 67.7 [48.6 to 83.3]

19. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With ≥0.5 log10 Change From Day 8 Baseline to Week 97 in HIV-1 RNA
Description: The percentage of participants in the pooled treatment group with ≥0.5 log10 change from baseline Day 8 to Week 97 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 8 (baseline) and Week 97
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 26
Percentage of participants | 69.2 [48.2 to 85.7]

20. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With ≥1.0 log10 Change From Day 1 Baseline to Week 25 in HIV-1 RNA
Description: The percentage of participants in the pooled treatment group with ≥1.0 log10 change from baseline Day 1 to Week 25 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 1 (baseline) and Week 25
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 34
Percentage of participants | 67.6 [49.5 to 82.6]

21. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With ≥1.0 log10 Change From Day 1 Baseline to Week 49 in HIV-1 RNA
Description: The percentage of participants in the pooled treatment group with ≥1.0 log10 change from baseline Day 1 to Week 49 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 1 (baseline) and Week 49
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 31
Percentage of participants | 71.0 [52.0 to 85.8]

22. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With ≥1.0 log10 Change From Day 1 Baseline to Week 97 in HIV-1 RNA
Description: The percentage of participants in the pooled treatment group with ≥1.0 log10 change from baseline Day 1 to Week 97 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 1 (baseline) and Week 97
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 26
Percentage of participants | 73.1 [52.2 to 88.4]

23. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With ≥1.0 log10 Change From Day 8 Baseline to Week 25 in HIV-1 RNA
Description: The percentage of participants in the pooled treatment group with ≥1.0 log10 change from baseline Day 8 to Week 25 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 8 (baseline) and Week 25
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 34
Percentage of participants | 58.8 [40.7 to 75.4]

24. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With ≥1.0 log10 Change From Day 8 Baseline to Week 49 in HIV-1 RNA
Description: The percentage of participants in the pooled treatment group with ≥1.0 log10 change from baseline Day 8 to Week 49 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 8 (baseline) and Week 49
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 31
Percentage of participants | 61.3 [42.2 to 78.2]

25. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With ≥1.0 log10 Change From Day 8 Baseline to Week 97 in HIV-1 RNA
Description: The percentage of participants in the pooled treatment group with ≥1.0 log10 change from baseline Day 8 to Week 97 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 8 (baseline) and Week 97
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 26
Percentage of participants | 61.5 [40.6 to 79.8]

26. Secondary Outcome: Mean Change From Baseline Day 1 to Week 25 in HIV-1 RNA From the Pooled Treatment Group
Description: The change from baseline Day 1 to Week 25 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% confidence intervals (CIs) were calculated based on the t-distribution. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 1 (baseline) and Week 25
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: Log10 Copies/mL
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 34
Log10 Copies/mL | -1.89 [-2.33 to -1.45]

27. Secondary Outcome: Mean Change From Baseline Day 1 to Week 49 in HIV-1 RNA From the Pooled Treatment Group
Description: The change from baseline Day 1 to Week 49 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% confidence intervals (CIs) were calculated based on the t-distribution. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 1 (baseline) and Week 49
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: Log10 Copies/mL
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 31
Log10 Copies/mL | -2.00 [-2.47 to -1.53]

28. Secondary Outcome: Mean Change From Baseline Day 1 to Week 97 in HIV-1 RNA From the Pooled Treatment Group
Description: The change from baseline Day 1 to Week 97 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% confidence intervals (CIs) were calculated based on the t-distribution. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 1 (baseline) and Week 97
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: Log10 Copies/mL
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 26
Log10 Copies/mL | -2.01 [-2.51 to -1.52]

29. Secondary Outcome: Mean Change From Baseline Day 8 to Week 25 in HIV-1 RNA From the Pooled Treatment Group
Description: The change from baseline Day 8 to Week 25 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% confidence intervals (CIs) were calculated based on the t-distribution. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 8 (baseline) and Week 25
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: Log10 Copies/mL
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 34
Log10 Copies/mL | -1.16 [-1.56 to -0.77]

30. Secondary Outcome: Mean Change From Baseline Day 8 to Week 49 in HIV-1 RNA From the Pooled Treatment Group
Description: The change from baseline Day 8 to Week 49 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% confidence intervals (CIs) were calculated based on the t-distribution. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 8 (baseline) and Week 49
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: Log10 Copies/mL
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 31
Log10 Copies/mL | -1.32 [-1.72 to -0.91]

31. Secondary Outcome: Mean Change From Baseline Day 8 to Week 97 in HIV-1 RNA From the Pooled Treatment Group
Description: The change from baseline Day 8 to Week 97 in HIV-1 RNA was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% confidence intervals (CIs) were calculated based on the t-distribution. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 8 (baseline) and Week 97
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: Log10 Copies/mL
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 26
Log10 Copies/mL | -1.36 [-1.83 to -0.89]

32. Secondary Outcome: Percentage of Participants From Day 1 Baseline to Day 8 With HIV-1 RNA <200 Copies mL
Description: The percentage of participants with HIV-1 RNA <200 copies mL was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% CIs were calculated based on the Clopper-Pearson method.
Time Frame: Day 1 (baseline) and Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 7 | 7
Percentage of participants
  Day 1 | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 41.0]
  Day 8 | 0.0 [0.0 to 41.0] | 14.3 [1.8 to 42.8] | 14.3 [0.4 to 57.9] | 0.0 [0.0 to 41.0]

33. Secondary Outcome: Percentage of Participants From Day 1 Baseline to Day 8 With HIV-1 RNA <50 Copies mL
Description: The percentage of participants with HIV-1 RNA <50 copies mL was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% CIs were calculated based on the Clopper-Pearson method.
Time Frame: Day 1 (baseline) and Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 7 | 7
Percentage of participants
  Day 1 | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 41.0]
  Day 8 | 0.0 [0.0 to 41.0] | 14.3 [1.8 to 42.8] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 41.0]

34. Secondary Outcome: Percentage of Participants From Day 1 Baseline to Day 8 With HIV-1 RNA <40 Copies mL
Description: The percentage of participants with HIV-1 RNA <40 copies mL was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% CIs were calculated based on the Clopper-Pearson method.
Time Frame: Day 1 (baseline) and Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ISL + ART | DOR + ART | DOR/ISL + ART | Placebo + ART
Number analyzed (Participants) | 7 | 14 | 7 | 7
Percentage of participants
  Day 1 | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 41.0]
  Day 8 | 0.0 [0.0 to 41.0] | 14.3 [1.8 to 42.8] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 41.0]

35. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With HIV-1 RNA <200 Copies/mL at Week 25
Description: The percentage of participants with HIV-1 RNA <200 copies mL at week 25 was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% CIs were calculated based on the Clopper-Pearson method. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Week 25
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 34
Percentage of participants | 64.7 [46.5 to 80.3]

36. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With HIV-1 RNA <200 Copies/mL at Week 49
Description: The percentage of participants with HIV-1 RNA <200 copies mL at week 49 was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% CIs were calculated based on the Clopper-Pearson method. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Week 49
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 31
Percentage of participants | 77.4 [58.9 to 90.4]

37. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With HIV-1 RNA <200 Copies/mL at Week 97
Description: The percentage of participants with HIV-1 RNA <200 copies mL at week 97 was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% CIs were calculated based on the Clopper-Pearson method. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Week 97
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 26
Percentage of participants | 80.8 [60.6 to 93.4]

38. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With HIV-1 RNA <50 Copies/mL at Week 25
Description: The percentage of participants with HIV-1 RNA <50 copies mL at week 25 was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% CIs were calculated based on the Clopper-Pearson method. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Week 25
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 34
Percentage of participants | 58.8 [40.7 to 75.4]

39. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With HIV-1 RNA <50 Copies/mL at Week 49
Description: The percentage of participants with HIV-1 RNA <50 copies mL at week 49 was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% CIs were calculated based on the Clopper-Pearson method. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Week 49
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 31
Percentage of participants | 71.0 [52.0 to 85.8]

40. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With HIV-1 RNA <50 Copies/mL at Week 97
Description: The percentage of participants with HIV-1 RNA <50 copies mL at week 97 was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% CIs were calculated based on the Clopper-Pearson method. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Week 97
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 26
Percentage of participants | 69.2 [48.2 to 85.7]

41. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With HIV-1 RNA <40 Copies/mL at Week 25
Description: The percentage of participants with HIV-1 RNA <40 copies mL at week 25 was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% CIs were calculated based on the Clopper-Pearson method. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Week 25
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 34
Percentage of participants | 58.8 [40.7 to 75.4]

42. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With HIV-1 RNA <40 Copies/mL at Week 49
Description: The percentage of participants with HIV-1 RNA <40 copies mL at week 49 was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% CIs were calculated based on the Clopper-Pearson method. Analysis of the pooled treatment group was planned per protocol.
Time Frame: Week 49
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 31
Percentage of participants | 71.0 [52.0 to 85.8]

43. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With HIV-1 RNA <40 Copies/mL at Week 97
Description: The percentage of participants with HIV-1 RNA <40 copies mL at week 97 was determined by the central laboratory using an Abbott Real Time PCR assay with a LLOD of 40 copies/mL. The within-group 95% CIs were calculated based on the Clopper-Pearson method. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Week 97
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 26
Percentage of participants | 69.2 [48.2 to 85.7]

44. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With Treatment-emergent Resistance-associated Substitutions to DOR at Week 25
Description: The prevalence of viral drug resistance to DOR was based on the percentage of participants with treatment-emergent (TE) resistance-associated substitutions (RASs), which is calculated by dividing the number of participants with TE RASs by the number of participants tested for resistance multiplied by 100. RASs for DOR were as follows: V106A/M, Y188C/L, F227C/H/I/L, M230I/L, L234I, Y318F, V108I, Y188F/H, G190E, H221Y, P236, and were determined by the central laboratory with the GenoSure Prime assay on post randomization samples from participants with HIV-1 RNA ≥200 copies/mL Analysis of the pooled treatment group was planned per protocol.
Time Frame: Week 25
Population: Randomized participants who received at least 1 dose of study intervention, had HIV-1 RNA ≥200 copies/mL, and were tested for resistance.
Measure: Number; unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 12
Percentage of participants | 33.3

45. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With Treatment-emergent Resistance-associated Substitutions to DOR at Week 49
Description: The prevalence of viral drug resistance to DOR was based on the percentage of participants with TE RASs, which is calculated by dividing the number of participants with TE RASs by the number of participants tested for resistance, multiplied by 100. RASs for DOR were as follows: V106A/M, Y188C/L, F227C/H/I/L, M230I/L, L234I, Y318F, V108I, Y188F/H, G190E, H221Y, P236, and were determined by the central laboratory with the GenoSure Prime assay on post randomization samples from participants with HIV-1 RNA ≥200 copies/mL Analysis of the pooled treatment group was planned per protocol.
Time Frame: Week 49
Population: as for outcome 44
Measure: Number; unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 7
Percentage of participants | 28.6

46. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With Treatment-emergent Resistance-associated Substitutions to ISL at Week 25
Description: The prevalence of viral drug resistance to ISL was based on the percentage of participants with TE RAS, which is calculated by dividing the number of participants with TE RAS by the number of participants tested for resistance, multiplied by 100. The RAS for ISL, M184V was determined by the central laboratory with the GenoSure Prime assay on post randomization samples from participants with HIV-1 RNA ≥200 copies/mL Analysis of the pooled treatment group was planned per protocol.
Time Frame: Week 25
Population: as for outcome 44
Measure: Number; unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 12
Percentage of participants | 8.3

47. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With Treatment-emergent Resistance-associated Substitutions to ISL at Week 49
Description: as for outcome 46
Time Frame: Week 49
Population: as for outcome 44
Measure: Number; unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 7
Percentage of participants | 14.3

48. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With Treatment-emergent Resistance-associated Substitutions to Optimized Background Therapy (OBT) Components at Week 25
Description: The prevalence of viral drug resistance to OBT components was based on the percentage of participants with TE RASs, which is calculated by dividing the number of participants with TE RASs by the number of participants tested for resistance, multiplied by 100. The RASs for OBT components were determined by the central laboratory with the GenoSure Prime assay on post randomization samples from participants with HIV-1 RNA ≥200 copies/mL Analysis of the pooled treatment group was planned per protocol.
Time Frame: Week 25
Population: as for outcome 44
Measure: Number; unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 12
Percentage of participants | 25.0

49. Secondary Outcome: Percentage of Participants From the Pooled Treatment Group With Treatment-emergent Resistance-associated Substitutions to OBT Components at Week 49
Description: as for outcome 48
Time Frame: Week 49
Population: as for outcome 44
Measure: Number; unit: Percentage of participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 7
Percentage of participants | 28.6

50. Secondary Outcome: Number of Participants From the Pooled Treatment Group With Viral Resistance-associated Substitutions (RASs) at Week 25
Description: The number of participants from the pooled treatment group who had HIV-1 RNA ≥200 copies/mL with treatment emergent RAS at week 25 showing the type of RAS .Analysis of the pooled treatment group was planned per protocol,
Time Frame: Week 25
Population: All randomized participants who received at least 1 dose of study intervention and had baseline data for those analyses that require baseline data. with confirmed HIV-1 RNA 200 copies/mL, and with available genotypic or phenotypic data that show evidence of resistance irrespective of viral load.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 12
Participants
  RAS A98G | 2
  RAS D67N | 1
  RAS H221Y | 1
  RAS K103S | 1
  RAS K219E | 1
  RAS L234I | 1
  RAS M184V | 1
  RAS M41L | 1
  RAS N348I | 1
  RAS V106A | 3
  RAS V106I | 2
  RAS V106M | 1
  RAS V179I | 2
  RAS Y318F | 1
  RAS F53L | 1
  RAS L90M | 1
  RAS M36I | 1

51. Secondary Outcome: Number of Participants From the Pooled Treatment Group With Viral RASs at Week 49
Description: The number of participants from the pooled treatment group who had HIV-1 RNA ≥200 copies/mL with treatment emergent RAS at week 49 showing the type of RAS .Analysis of the pooled treatment group was planned per protocol,
Time Frame: Week 49
Population: All randomized participants who received at least 1 dose of study intervention and had baseline data for those analyses that require baseline data. with confirmed HIV-1 RNA ≥200 copies/mL, and with available genotypic or phenotypic data that show evidence of resistance irrespective of viral load.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 7
Participants
  RAS A98G | 1
  RAS D67N | 1
  RAS K103S | 1
  RAS K219E | 1
  RAS M184V | 1
  RAS M41L | 1
  RAS N348I | 1
  RAS V106A | 2
  RAS V106I | 1
  RAS V106M | 1
  RAS V179I | 2
  RAS F53L | 1
  RAS L90M | 1
  RAS M36I | 1

52. Secondary Outcome: Number of Participants From the Pooled Treatment Group With Viral RASs at Week 97
Description: The number of participants from the pooled treatment group with treatment emergent RAS at week 97 are presented, showing the type of RAS .Analysis of the pooled treatment group was planned per protocol,
Time Frame: Week 97
Population: All randomized participants who received at least 1 dose of study intervention and had baseline data for those analyses that require baseline data. with confirmed HIV-1 RNA ≥400 copies/mL, and with available genotypic or phenotypic data that show evidence of resistance irrespective of viral load.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 5
Participants
  RAS D67N | 1
  RAS M41L | 1
  RAS N348I | 1
  RAS T215F | 1
  RAS V106A | 2
  RAS V106I | 1
  RAS V106M | 1
  RAS V179I | 1
  RAS F53L | 1
  RAS L90M | 1
  RAS M36I | 1

53. Secondary Outcome: Number of Participants From the Pooled Treatment Group Exhibiting Antiviral Resistance of HIV-1 RNA ≥200 Copies/mL at Week 25
Description: The number of participants from the pooled treatment group exhibiting antiviral resistance of HIV-1 RNA ≥200 copies/mL at Week 25 is presented. .Analysis of the pooled treatment group was planned per protocol,
Time Frame: Week 25
Population: as for outcome 52
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 35
Participants | 12

54. Secondary Outcome: Number of Participants From the Pooled Treatment Group Exhibiting Antiviral Resistance of HIV-1 RNA ≥200 Copies/mL at Week 49
Description: The number of participants from the pooled treatment group exhibiting antiviral resistance of HIV-1 RNA ≥200 copies/mL at Week 49 is presented. .Analysis of the pooled treatment group was planned per protocol,
Time Frame: Week 49
Population: as for outcome 52
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 35
Participants | 7

55. Secondary Outcome: Number of Participants From the Pooled Treatment Group Exhibiting Antiviral Resistance of HIV-1 RNA ≥200 Copies/mL at Week 97
Description: The number of participants from the pooled treatment group exhibiting antiviral resistance of HIV-1 RNA ≥200 copies/mL at Week 97 is presented. .Analysis of the pooled treatment group was planned per protocol,
Time Frame: Week 97
Population: as for outcome 52
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 35
Participants | 5

56. Secondary Outcome: Change From Baseline Day 1 to Week 25 in Cluster of Differentiation 4+ (CD4+) T-cell Counts From the Pooled Treatment Group
Description: The change from baseline Day 1 to Week 25 in CD4+ T-cell counts was determined by the central laboratory.. The within-group 95% CIs were calculated based on the t-distribution. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 1 (baseline) and Week 25
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 30
cells/mm^3 | 50.3 [27.8 to 72.9]

57. Secondary Outcome: Change From Baseline Day 1 to Week 49 in CD4+ T-cell Counts From the Pooled Treatment Group
Description: The change from baseline Day 1 to Week 49 in CD4+ T-cell counts was determined by the central laboratory.. The within-group 95% CIs were calculated based on the t-distribution. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 1 (baseline) and Week 49
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 30
cells/mm^3 | 86.9 [51.2 to 122.5]

58. Secondary Outcome: Change From Baseline Day 1 to Week 97 in CD4+ T-cell Counts From the Pooled Treatment Group
Description: The change from baseline Day 1 to Week 97 in CD4+ T-cell counts was determined by the central laboratory.. The within-group 95% CIs were calculated based on the t-distribution. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 1 (baseline) and Week 97
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 24
cells/mm^3 | 114.6 [54.7 to 174.6]

59. Secondary Outcome: Change From Baseline Day 8 to Week 25 in CD4+ T-cell Counts From the Pooled Treatment Group
Description: The change from baseline Day 8 to Week 25 in CD4+ T-cell counts was determined by the central laboratory.. The within-group 95% CIs were calculated based on the t-distribution. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 8 (baseline) and Week 25
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 30
cells/mm^3 | 38.0 [9.6 to 66.4]

60. Secondary Outcome: Change From Baseline Day 8 to Week 49 in CD4+ T-cell Counts From the Pooled Treatment Group
Description: The change from baseline Day 8 to Week 49 in CD4+ T-cell counts was determined by the central laboratory.. The within-group 95% CIs were calculated based on the t-distribution. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 8 (baseline) and Week 49
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 30
cells/mm^3 | 75.1 [36.9 to 113.4]

61. Secondary Outcome: Change From Baseline Day 8 to Week 97 in CD4+ T-cell Counts From the Pooled Treatment Group
Description: The change from baseline Day 8 to Week 97 in CD4+ T-cell counts was determined by the central laboratory.. The within-group 95% CIs were calculated based on the t-distribution. Analysis of the pooled treatment group was planned per protocol,
Time Frame: Day 8 (baseline) and Week 97
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Pooled Treatment
Number analyzed (Participants) | 24
cells/mm^3 | 108.0 [47.9 to 168.2]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality (ACM): from randomization up to Week 49; Adverse Events (AE): from treatment ( Day 1) Up to Week 97
Description: All randomized participants who received at least 1 dose of study intervention based on the treatment group to which they were randomized.
Groups:
- ISL+ART: HTE participants with HIV-1 infection took islatravir (ISL) 0.75 mg once daily (QD) in combination with failing ART from Day 1 to Day 7; followed by open-label 100 mg doravirine (DOR)/0.75 mg ISL fixed dose combination (FDC) QD + optimized background therapy (OBT) from Day 8 to Week 97.
- DOR+ART: HTE participants with HIV-1 infection took DOR 100 mg QD in combination with failing ART from Day 1 to Day 7; followed by open-label 100 mg DOR/0.75 mg ISL FDC QD + OBT from Day 8 to Week 97.
- DOR/ISL+ART: HTE participants with HIV-1 infection took 100 mg DOR/0.75 mg ISL FDC QD in combination with failing ART from Day 1 to Day 7; followed by open-label 100 mg DOR/0.75 mg ISL FDC QD + OBT from Day 8 to Week 97.
- Placebo+ART: HTE participants with HIV-1 infection took placebo QD in combination with failing ART from Day 1 to Day 7; followed by open-label 100 mg DOR/0.75 mg ISL FDC QD + OBT from Day 8 to Week 97.
Arm/Group | ISL+ART | DOR+ART | DOR/ISL+ART | Placebo+ART
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/14 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7 | 2/14 | 0/7 | 2/7
Other Adverse Events (participants affected / at risk) | 6/7 | 14/14 | 6/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISL+ART (N=7) | DOR+ART (N=14) | DOR/ISL+ART (N=7) | Placebo+ART (N=7)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SARS-CoV-2 sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reactive gastropathy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISL+ART (N=7) | DOR+ART (N=14) | DOR/ISL+ART (N=7) | Placebo+ART (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye allergy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal rash (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (5) | 2 (3) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (2) | 1 (1) | 1 (1) | 2 (2)
Exercise tolerance decreased (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Amoebiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal foot infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (4) | 1 (3) | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal transit time increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 5 (6) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep terror (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturnal hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT04233216/Prot_SAP_000.pdf